CLINICAL TRIAL: NCT00276250
Title: Development of Immunosuppression Regimens to Facilitate Single Donor Islet Transplantation Using Abatacept
Brief Title: Islet Transplantation Using Abatacept
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Nicole Turgeon MD, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00021852; 1136-2005 (Other: Emory University)
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Results first posted 2016-07-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-06

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — efalizumab; Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Efalizumab Followed by Abatacept Regimen (Experimental): Participants with Type 1 diabetes with onset of disease at < 40 years of age and insulin-dependence for > 5 years received efalizumab-based immunosuppression regimen after islet-cell transplantation. During the course of the study, efalizumab was withdrawn from the US market due to safety concerns. The protocol was subsequently amended to alter the immunosuppressive regimen to abatacept for these participants.
  Interventions: Drug: Efalizumab; Drug: Abatacept
- Abatacept Regimen (Experimental): Participants with Type 1 diabetes with onset of disease at < 40 years of age and insulin-dependence for > 5 years received abatacept immunosuppresion regimen after islet-cell transplantation.
  Interventions: Drug: Abatacept
- Belatacept Regimen (Experimental): Participants with Type 1 diabetes with onset of disease at < 40 years of age and insulin-dependence for > 5 years received Belatacept immunosuppresion regimen after islet-cell transplantation.
  Interventions: Drug: Belatacept

INTERVENTIONS:
Drug: Efalizumab — Efalizumab was a medication approved for use in psoriasis which was being explored to determine efficacy with immunosuppression following organ transplantation. Efalizumab was administered subcutaneously on a weekly basis. Upon efalizumab being withdrawn from the US market, the protocol was amended to alter the immunosuppressive regimen to abatacept for the study participants.
  Other Names: Raptiva
  Arms: Efalizumab Followed by Abatacept Regimen
Drug: Abatacept — Abatacept is drug used to treat autoimmune diseases. Abatacept is administered intravenously, monthly, in weight-based doses and is given for as long as transplanted islets are functioning.
  Other Names: Orencia
  Arms: Abatacept Regimen; Efalizumab Followed by Abatacept Regimen
Drug: Belatacept — Belatacept is a medication to provide extended graft survival while limiting the toxicity generated by standard immune suppressing regimens. Belatacept is administered intravenously. The protocol for this study was amended to substitute belatacept for abatacept for all newly enrolling participants (current participants remained on abatacept).
  Other Names: Nulojix
  Arms: Belatacept Regimen

SUMMARY:
Islet transplantation in type 1 diabetics with hypoglycemic unawareness using abatacept as a part of a novel calcineurin-inhibitor-sparing immunosuppressive regimen.

DETAILED DESCRIPTION:
More than 1 million North Americans have type 1 diabetes. Each year, approximately 30,000 new cases of type 1 diabetes are diagnosed in the United States. Type 1 diabetes destroys islets, a cluster of cells within the pancreas that produce insulin. Insulin is a hormone with many effects. However, the most important effect of insulin is to control the level of sugar in the blood. People with Type 1 diabetes no longer produce insulin and must take insulin injections to live. Despite steady improvements in the management of this disease, its victims remain at increased risk for stroke, heart attack, kidney failure, amputation, blindness, nerve damage and premature death. The life expectancy of a teenager is reduced by thirty years from the time of onset of the disease [1]. Unfortunately, many type 1 diabetics cannot control their blood sugars in spite of very careful monitoring and the frequent injection of insulin. This group of patients is considered to have labile or "brittle" diabetes. These "brittle" diabetics can often have wide swings in their blood sugar levels that can be life threatening. Hypoglycemia, or low blood sugars occur when too much insulin is in the bloodstream. When this occurs, it is vital that patients eat or drink something right away that will increase their blood sugars. Many diabetics lose the ability to recognize when their blood sugars are getting dangerously low. These episodes of hypoglycemia can lead to coma, and possibly death, if not recognized and treated right away. Patients can also experience extreme increases in blood sugars, or hyperglycemia, as a result of emotional or physical stress. Hyperglycemia can result in dehydration, confusion, and a condition called ketoacidosis, which can lead to death. When this happens, insulin must be given as soon as possible.

Islet transplantation can restore the body's ability to make insulin and, in turn, restore normal blood sugar levels.

Since the 1960's, doctors and scientists have attempted to replace this islet function by performing whole organ pancreas transplantation. While the results of pancreas transplantation have improved dramatically in recent years, this approach has largely been limited to patients with kidney disease who have also needed a kidney transplant. This is because of the risks associated with the surgical procedure and the immunosuppressive drugs required to prevent rejection or the destruction of the transplanted pancreas by the body's immune system [2]. Transplantation of a whole pancreas requires a major operation that is done through an incision in the abdomen. The patient must be under general anesthesia, or asleep, for the entire procedure. Recent clinical experience suggests that islet transplantation may be a useful approach to correct diabetes in humans [3].

Islet transplantation offers a direct approach to the treatment of type 1 diabetes. A large number of experimental studies carried out in many laboratories over the last decade have documented the beneficial effects of islet transplants in experimental animals. These experiments have confirmed both the efficiency and safety of islet transplantation [4,5].

The inability to isolate enough islets from a single pancreas has been one obstacle to successful islet transplantation. A certain number of islets must be isolated, or separated, from a single pancreas in order to use them for transplant. If this minimum number of islets is not obtained, then the islets do not effectively reverse diabetes. Progress in isolating the islets from a human pancreas has been dramatic in the last several years. Advances in equipment and technology have lead to increases in the number of islets that can be isolated from a single pancreas.

After successful isolation, the islets can be injected through a catheter into the patient's liver during a thirty-minute procedure. A group of doctors at the University of Alberta in Edmonton, Canada has had promising results in human islet transplantation. Normal sugar levels have been documented after human islet transplants. Also, recent improvements in immunosuppressive drug treatments have resulted in sustained insulin-independence in selected type 1 diabetic patients [6-9,10,11,12]. The traditional method of transplant immunosuppression includes using some form of a steroid drug. Steroids have been found to injure or kill the islets after transplant. The doctors in Edmonton, Canada established an immunosuppression formula that does not use steroids. The objective of the study here at Emory University is to reproduce the successful results of human islet transplantation that have been achieved by the doctors at the University of Alberta using steroid free immunosuppression.

The Emory Islet Transplant Program will enroll up to 20 participants, ages 18 to 65, in this study. Each of the twenty patients will receive up to 3 islet infusions from three different cadaver donors. Each patient will be placed on immunosuppressive drugs to prevent the body from rejecting or destroying the transplanted islets. In this study we are using a medication, abatacept, to help prevent organ rejection. This medication has been previously used in people to treat psoriasis. The participants will also receive basiliximab and sirolimus as immunosuppressant medications.

Each patient will have his/her blood sugar levels and insulin requirements monitored very closely after each transplant. The patients will also have various tests to determine if their diabetic complications improve, remain the same, or become worse. The patients will be asked to record any episodes of hypoglycemia or low blood sugars while participating in this study. Emory will examine whether or not there is a decrease in how often the episodes occur. Patients will also undergo regular eye exams to document retinal changes or improvements that may occur after transplant. At this time it is not known whether islet transplantation slows or stops the progression of common diabetic complications. More experience and research is needed before this can be determined. One focus of our research will be to study diabetic complications in patients who receive islet transplants.

The major goal of the Emory Islet Transplant Program is for patients participating in this study to be free of the need for insulin injections after 2 islet transplants. Because many advances have been made in islet transplantation, the transplant team at Emory would like to participate in this promising treatment of type 1 diabetes and, most importantly, help those who suffer from this disease become free from daily insulin injections and avoid the devastating complications that happen as a result of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients age 18 to 65 years of age
* Clinical history compatible with type 1 diabetes with onset of disease at <40 years of age and insulin-dependence for >5 years at the time of enrollment.
* Body mass index less than or equal to 26
* 18 to 65 years of age
* Absent stimulated C-peptide (<0.3ng/ml) in response to a mixed meal tolerance test (Boost® 6 mL/kg body weight to a maximum of 360 mL; another product with equivalent caloric and nutrient content may be substituted for Boost) measured at 90min after the end of consumption.
* Compliance with an optimized diabetic management plan as assessed by an Emory University endocrinologist
* Checking and recording blood sugars at least 3 times per day
* Involvement in intensive diabetes management defined as self monitoring of glucose values no less than a mean of three times each day averaged over each week and by the administration of three or more insulin injections each day or insulin pump therapy. Such management must be under the direction of an endocrinologist, diabetologist, or diabetes specialist with at least 3 clinical evaluations during the previous 12 months.
* At least one episode of severe hypoglycemia in the past 3 years defined as an event with symptoms compatible with hypoglycemia in which the subject required the assistance of another person and which was associated with either a blood glucose level <50 mg/dL [2.8 mmol/L] or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration).
* Reduced awareness of hypoglycemia as defined by a Clarke score of 4 or more and a HYPO score greater than or equal to the 90th percentile (1047) within the last 6 months prior to randomization; OR Marked glycemic lability characterized by wide swings in blood glucose despite optimal diabetes therapy and defined by a glycemic lability index (LI) score greater than or equal to the 90th percentile (433 mM2/h/wk) within the last 6 months prior to randomization; OR A composite of a Clarke score of 4 or more and a HYPO score greater than or equal to the 75th percentile (423) and a LI greater than of equal to the 75th percentile (329) within the last 6 months prior to randomization.

Exclusion Criteria:

* Severe co-existing cardiac disease, characterized by any one of these conditions:
* Recent myocardial infarction (within past six months)
* Left Ventricular Ejection Fraction < 30%
* Evidence of ischemia on a functional echocardiogram
* Active infection including hepatitis B, hepatitis C, HIV, or TB as determined by a positive skin test or clinical presentation, or under treatment for suspected TB. Positive tests are acceptable only if associated with a history of previous vaccination in the absence of any sign of active infection. Positive tests are otherwise not acceptable, even in the absence of any active infection at the time of evaluation
* Invasive aspergillus infection within one year prior to study entry.
* Negative screen for Epstein-Barr Virus (EBV) by IgG determination.
* Administration of live vaccine within the past two months
* Measured glomerular filtration rate using iohexol <70 mL/min/1.73 m2 for females and <80 mL/min/1.73 m2 for males (or a 24 hr. creatinine clearance with participants allergic to iodine <85mL/min/1.73m2).
* Macroalbuminuria (urinary protein excretion rate >300 mg/24h)
* Baseline Hgb below the lower limits of normal at the local laboratory; lymphopenia (<1,000/L), neutropenia (<1,500/L), or thrombocytopenia (platelets <100,000/ L).
* Hyperlipidemia (fasting LDL cholesterol >130 mg/dL, treated or untreated; and/or fasting triglycerides >300 mg/dL)
* Negative antibody test for Varicella zoster virus (subjects may be reconsidered if they receive the vaccination and convert to a positive antibody)
* History of malignancy (except squamous or basal cell skin carcinoma) within the previous 5 years
* Previous/concurrent organ transplantation
* Presence of HLA Panel Reactive Antibodies >20%
* Active peptic ulcer disease
* Evidence of gallbladder disease including cholecystitis and cholelithiasis
* Evidence of liver disease including: hepatic neoplasm, portal hypertension, or persistently abnormal liver function tests
* Current use of systemic steroid medications
* Evidence of insulin resistance (insulin requirements >0.8 units/kg/day)
* Inability to provide informed consent
* Severe unremitting diarrhea, vomiting or other gastrointestinal disorders potentially interfering with the ability to absorb oral medications.
* Hyperlipidemia despite medical therapy (fasting LDL cholesterol >130 mg/dL, treated or untreated; and/or fasting triglycerides >200 mg/dL).
* Acute or chronic pancreatitis.
* Symptomatic peptic ulcer disease.
* Use of any other investigational agents within 4 weeks of participation.
* Any condition or any circumstance that makes it unsafe to undergo an islet cell transplant
* Any coagulopathy or medical condition requiring long-term anticoagulant therapy (e.g., warfarin) after transplantation (low-dose aspirin treatment is allowed) or patients with an INR >1.5.
* Sickle Cell Anemia (Subjects with Sickle Cell Anemia, trait HbSS, are at high risk for complications after transplantation related to immunosuppressive therapy. These complications include stroke and sickle cell crisis. Therefore, we will exclude these subjects from our study to minimize risks to study subjects.)
* For female participants: Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study and 3 months after discontinuation. For male participants: intent to procreate during the duration of the study or within 3 months after discontinuation or unwillingness to use effective measures of contraception. Oral contraceptives, Norplant®, Depo-Provera®, and barrier devices with spermicide are acceptable contraceptive methods; condoms used alone are not acceptable.
* Active alcohol or substance abuse. This includes cigarette smoking (must be abstinent for six months). Active alcohol abuse should be considered using the current NIAAA definitions, whereby alcohol abuse is defined by a pattern of drinking that is accompanied by one or more of the following situations within a 12-month period:
* Failure to fulfill major work, school, or home responsibilities
* Drinking in situations that are physically dangerous, such as while driving a car or operating machinery
* Recurring alcohol-related legal problems, such as driving under the influence of alcohol or for causing physical harm to someone while intoxicated
* Continued alcohol abuse despite having ongoing relationship problems that are caused or worsened by the effects of alcohol
* Psychiatric disorder making the subject not a suitable candidate for transplantation, e.g., schizophrenia, bipolar disorder, or major depression that is unstable or uncontrolled on current medication. (A psychological or psychiatric consultation is required only if considered necessary by some current indication or history.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2005-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian P Larsen, MD, D.Phil, Principal Investigator — Emory University; Thomas C Pearson, MD, D,Phil, Principal Investigator — Emory University; Sallie C Carpentier, RN, BSN, Study Director — Emory University; Nicole Turgeon, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Nine subjects signed informed consent. During evaluation, four participants were found ineligible for study inclusion. Five participants completed the evaluation process and were listed for an islet transplant
Period: Overall Study
Arm/Group | Efalizumab Followed by Abatacept Regimen | Abatacept Regimen | Belatacept Regimen
Started | 4 | 1 | 0
Completed | 4 | 1 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Efalizumab Followed by Abatacept Regimen | Abatacept Regimen | Belatacept Regimen | Total
Number analyzed (Participants) | 4 | 1 | 0 | 5
Age, Categorical [Number; unit: participants]
  <=18 years | 0 | 0 |  | 0
  Between 18 and 65 years | 4 | 1 |  | 5
  >=65 years | 0 | 0 |  | 0
Gender [Number; unit: participants]
  Female | 1 | 1 |  | 2
  Male | 3 | 0 |  | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 | 1 |  | 5

OUTCOME MEASURES:

1. Primary Outcome: The Number of Insulin-independent Subjects at Day 75 (± 5 Days) Following the First Islet Cell Transplantation
Time Frame: 75 days post-transplantation
Measure: Number; unit: participants
Arm/Group | Efalizumab Followed by Abatacept Regimen | Abatacept Regimen | Belatacept Regimen
Number analyzed (Participants) | 4 | 1 | 0
participants | 4 | 1 |

2. Secondary Outcome: Number of Insulin-independent Subjects Following Islet Transplantation
Description: Participants who did not need to take insulin at 1, 3, 6, 9, 12, 18, and 24 months following islet transplantation
Time Frame: 1, 3, 6, 9,12,18 and 24 months post-transplantation
Measure: Number; unit: participants
Arm/Group | Efalizumab Followed by Abatacept Regimen | Abatacept Regimen | Belatacept Regimen
Number analyzed (Participants) | 4 | 1 | 0
participants
  1 Month Post-Transplant | 4 | 0 |
  3 Months Post-Transplant | 4 | 0 |
  6 Months Post-Transplant | 4 | 0 |
  9 Months Post-Transplant | 3 | 0 |
  12 Months Post-Transplant | 3 | 0 |
  18 Months Post-Transplant | 2 | 0 |
  24 Months Post-Transplant | 2 | 0 |

3. Secondary Outcome: Number of Subjects With HbA1C Less Than 6.5%
Description: HbA1C was assessed in the subjects 6 months after transplantation and the number of subjects with values less than 6.5% was recorded which indicated better control of blood glucose levels.
Time Frame: 6 months post-transplantation
Population: The HbA1C for the subject in the abatacept arm was above the threshold (6.5%) for this measure.
Measure: Number; unit: participants
Arm/Group | Efalizumab Followed by Abatacept Regimen | Abatacept Regimen | Belatacept Regimen
Number analyzed (Participants) | 4 | 1 | 0
participants | 4 | 0 |

4. Secondary Outcome: Number of Subjects With HbA1C Levels < 6.5%
Description: HbA1C was assessed in the subjects 12 months after transplantation and the number of subjects with levels < 6.5% was recorded which indicated better control of blood glucose levels.
Time Frame: 12 months post-transplantation
Measure: Number; unit: participants
Arm/Group | Efalizumab Followed by Abatacept Regimen | Abatacept Regimen | Belatacept Regimen
Number analyzed (Participants) | 4 | 1 | 0
participants | 3 | 0 |

5. Secondary Outcome: Number of Subjects With HbA1C < 6.5%
Description: HbA1C was assessed in the subjects 24 months after transplantation and the number of subjects with levels < 6.5% was recorded which indicated better control of blood glucose levels.
Time Frame: 24 months post-transplant
Population: One participant in the Efalizumab followed by abatacept regimen arm had partial graft function and withdrew from the study at 18 months post-transplantation (prior to this time point of assessment).
Measure: Number; unit: participants
Arm/Group | Efalizumab Followed by Abatacept Regimen | Abatacept Regimen | Belatacept Regimen
Number analyzed (Participants) | 3 | 1 | 0
participants | 2 | 0 |

6. Secondary Outcome: Number of Subjects With HbA1C < 6.5%
Description: HbA1C was assessed in the subjects 36 months after transplantation and the number of subjects with values < 6.5% was recorded which indicated better control of blood glucose levels.
Time Frame: 36 months post-transplantation
Population: Two participants in the Efalizumab followed by abatacept regimen arm were terminated prior to this time point due to islet graft failure; another one withdrew as they did not want to change to abatacept. The single participant in the Abatacept arm withdrew after graft failure which occurred at 6months post-transplantation.
Measure: Number; unit: participants
Arm/Group | Efalizumab Followed by Abatacept Regimen | Abatacept Regimen | Belatacept Regimen
Number analyzed (Participants) | 1 | 0 | 0
participants | 1 |  |

7. Secondary Outcome: Number of Participants With Endogenous Insulin Production Post-transplant, Assessed by Fasting C-peptide Levels
Description: The number of subjects exhibiting C-peptide levels ≥ 0.5 ng/mL was recorded.
Time Frame: 1, 3, 6, 9,12,18 and 24 months post-transplantation
Population: C-Peptide values were not obtained for 2 participants in the Efalizumab followed by abatacept arm at the 18 and 24 months post-transplant timepoints.
Measure: Number; unit: participants
Arm/Group | Efalizumab Followed by Abatacept Regimen | Abatacept Regimen | Belatacept Regimen
Number analyzed (Participants) | 4 | 1 | 0
participants
  1 Month Post-Transplant | 4 | 1 |
  3 Months Post-Transplant | 4 | 0 |
  6 Months Post-Transplant | 4 | 0 |
  9 Months Post-Transplant | 4 | 0 |
  12 Months Post-Transplant | 4 | 0 |
  18 Months Post-Transpla | 2 | 0 |
  24 Months Post-Transplant | 2 | 0 |

8. Secondary Outcome: The Number of Study Participants Exhibiting a Successful Response to a Standard Mixed Meal Test, Measured by Stimulated C-peptide Levels After Islet Transplant.
Description: The number of study participants who have detectable C-peptide levels after stimulation from a Mixed Meal Test. An increase of C-peptide indicates that insulin is being released normally in response to food consumption.
Time Frame: 1, 3, 6, 9,12,18 and 24 months post-transplantation
Population: C-Peptide values were not obtained for 2 participants in the Efalizumab followed by abatacept arm for 18 and 24 months post-transplant
Measure: Number; unit: participants
Arm/Group | Efalizumab Followed by Abatacept Regimen | Abatacept Regimen | Belatacept Regimen
Number analyzed (Participants) | 4 | 1 | 0
participants
  1 Month Post-Transplant | 4 | 0 |
  3 Months Post-Transplant | 4 | 0 |
  6 Months Post-Transplant | 4 | 0 |
  9 Months Post-Transplant | 3 | 0 |
  12 Months Post-Transplant | 3 | 0 |
  18 Months Post-Transpla | 2 | 0 |
  24 Months Post-Transplant | 2 | 0 |

9. Secondary Outcome: Number of Subjects With Normal Renal Function, as Measured by Serum Creatinine Levels
Description: Renal function was assessed by measuring levels of serum creatinine. Normal values range from 0.7 to 1.3 mg/dL for men and 0.6 to 1.1 mg/dL for women.
Time Frame: 24 months after transplant
Population: One subject in the Efalizumab followed by abatacept regimen arm withdrew from the the study at 18 months post-transplantation and therefore did not have the 24-month assessments.
Measure: Number; unit: participants
Arm/Group | Efalizumab Followed by Abatacept Regimen | Abatacept Regimen | Belatacept Regimen
Number analyzed (Participants) | 4 | 1 | 0
participants | 3 | 1 |

ADVERSE EVENTS:
Time Frame: Adverse events data will be collected from the point of islet transplantation throughout the duration of study participation, an average of 2 years.
Description: All adverse events will be recorded, regardless of the severity or relationship to study medication or procedure unless otherwise stated in the CIT-TCAE v. 3.0. Subjects experiencing adverse events will be treated appropriately and observed at suitable intervals until the events resolve or stabilize.
Arm/Group | Efalizumab Followed by Abatacept Regimen | Abatacept Regimen | Belatacept Regimen
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 4/4 | 1/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efalizumab Followed by Abatacept Regimen (N=4) | Abatacept Regimen (N=1) | Belatacept Regimen (N=0)
Fever with cough and chills (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — The participant was hospitalized over night and received IV antibiotics to treat an infection presenting with fever, cough and chills.
Vertigo (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — The participant was hospitalized for two days after experiencing vertigo that was progressing in severity. Diagnostic tests were all negative for acute neurological concerns and the participant was released from the hospital.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Efalizumab Followed by Abatacept Regimen (N=4) | Abatacept Regimen (N=1) | Belatacept Regimen (N=0)
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0
Elevated Liver Enzymes (Hepatobiliary disorders) | 2 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Increased Epstein-Barr Viral load assessed by Polymerase Chain Reaction (Infections and infestations) | 3 | 0 | 0

LIMITATIONS AND CAVEATS:
Enrollment in this study was limited by the removal of Efalizumab from the market in 2009 after patients (external to this study) being treated for plaque psoriasis were diagnosed with Progressive Multifocal Leukoencephalopathy (PML).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes